CLINICAL TRIAL: NCT02308696
Title: The Effectiveness of Peer-to-Peer Community Support to Promote Aging in Place
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Community Place (Unknown); Jewish Family Service of Los Angeles (Unknown); Alpert Jewish Family And Childrens Service (Other); Alliance for Children and Families (Unknown); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-1013; 000001 (Other: UW)
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Wellness Programs; Hospitalization; Emergency Room
Keywords: Older Adults; Aging in Place
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer-to-peer support (non-randomized) (Experimental): 225 older adults that are currently receiving peer-to-peer support
  Interventions: Behavioral: Peer-to-Peer Support
- Standard Services (non-randomized) (Active Comparator): 225 older adults will continue receiving standard community services
  Interventions: Behavioral: Standard Community Services

INTERVENTIONS:
Behavioral: Peer-to-Peer Support — All three data collection sites run peer-to-peer community support programs. Core program elements include the same program objective, standard definition of who qualifies for peer-to-peer support, the mechanism by which older adults are referred for consideration for peer-support, core elements of training programs for the older adults who volunteer to provide the peer support, and monthly in-service trainings for all volunteers once trained, weekly hours that volunteers spend providing support, and provision of small stipends for volunteers.As they find their role very rewarding, there is very little peer turn-over; the vast majority of peers volunteer for years in this role, until they themselves start requiring services.
  Arms: Peer-to-peer support (non-randomized)
Behavioral: Standard Community Services — All three data collection sites will continue to provide standard community services to the older adults that are not enrolled in the peer-to-peer support program
  Arms: Standard Services (non-randomized)

SUMMARY:
The investigators' overall objective is to evaluate the effectiveness of peer-to-peer support programs in preventing the necessity of acute health care and nursing home services for older adult populations and in promoting their health and wellness. The investigators' Specific Aims are:

1. To compare the effectiveness of peer-to-peer community support in preventing hospitalization, emergency department (ED) use, and nursing home placement in an at-risk older adult population relative to standard community services.
2. To compare the effect of peer-to-peer community support on intermediary measures of health and wellness such as self-rated health, depression, and anxiety relative to standard community services.

DETAILED DESCRIPTION:
The investigators will accomplish the aims by conducting a longitudinal comparative-effectiveness study in which at-risk older adult study participants in three communities across the US are followed for 12-months. Using a quasi-experimental design, investigators will compare outcomes in those receiving peer-to-peer community support to those receiving standard community services.

At all three sites investigators will include 120 older adults in the peer-to-peer support group and 120 in the standard community services group for a total intervention group size of 360 (120 from each site) and 360 in the control group (120 from each site).

Study Outcomes & Measures To meet the first two aims investigators will (1) compare annualized rates of hospitalization, ED use, and nursing home placement and (2) examine the changes in self-reported health, depression, anxiety, and other measures of well-being in the group receiving peer-to-peer support compared to the group receiving standard community services from baseline to the end of study enrolment. The investigators describe each of our outcomes and additional study measures in detail below. Measures have been translated and used in Spanish and have been shown to be valid or have high reliability in Spanish

ELIGIBILITY:
Inclusion Criteria:

* Overall

  * ≥65 years of age
  * Speaks English or Spanish
  * Lives independently in their community year-round
  * Meet the community defined criterion for receiving peer-to-peer support (at least one of the following)

    * Low income (at or below poverty level)
    * On a fixed income that barely meets their living expenses
    * Social and/or familial isolation
    * Chronic Illness
    * In need of frequent community services or resources. Peer-to-peer support group (must meet the overall inclusion criteria as well as the following)
  * Enrolled in the peer-to-peer support program and have an assigned peer volunteer

Exclusion Criteria:

* < 65
* Score ≤ 30 on the Telephone Interview of Cognitive Status (TICS) because they will not have the ability to complete the survey
* State that it is unlikely that they will receive peer-to-peer support services for at least a year. Individuals who are unlikely to receive at least a year of services include those who need short-term help after a surgery and are likely to return to full functioning and those planning to transition to nursing home care or move away.

  * Currently receiving hospice services

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 456 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Jacobs, MD MPP, Principal Investigator — UMadison
Locations (5):
- United States (5):
  - Jewish Family Service, Los Angeles, California
  - Alpert Jewish Family and Children's Service, West Palm Beach, Florida
  - Community Place of Greater Rochester, Rochester, New York
  - University of Wisconsin, Madison, Wisconsin
  - Aliance For Children and Families, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Peer-to-peer Support (Non-randomized): 222 older adults that are currently receiving peer-to-peer support
  Peer-to-Peer Support: All three data collection sites run peer-to-peer community support programs. Core program elements include the same program objective, standard definition of who qualifies for peer-to-peer support, the mechanism by which older adults are referred for consideration for peer-support, core elements of training programs for the older adults who volunteer to provide the peer support, and monthly in-service trainings for all volunteers once trained, weekly hours that volunteers spend providing support, and provision of small stipends for volunteers.As they find their role very rewarding, there is very little peer turn-over; the vast majority of peers volunteer for years in this role, until they themselves start requiring services.
- Standard Services (Non-randomized): 234 older adults will continue receiving standard community services
  Standard Community Services: All three data collection sites will continue to provide standard community services to the older adults that are not enrolled in the peer-to-peer support program
Period: Overall Study
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized)
Started | 222 | 234
Completed | 169 | 203
Not Completed | 53 | 31
Not completed — Lost to Follow-up | 28 | 21
Not completed — Death | 8 | 4
Not completed — Moved to a Higher Level of Care | 17 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized) | Total
Number analyzed (Participants) | 222 | 234 | 456
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 222 | 234 | 456
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 185 | 370
  Male | 37 | 49 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 24 | 25 | 49
  Asian | 2 | 2 | 4
  Hispanic | 21 | 24 | 45
  White | 173 | 183 | 356
  Other | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 222 | 234 | 456
Spanish Language Preferred [Count of Participants; unit: Participants] | 13 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Hospitalizations, Emergency Department Visits, and Urgent Care Visits
Description: Investigators will ask participants to report their hospitalizations, ED and Urgent Care visits over the course of a 1 year follow up
Time Frame: 1 year
Population: It was determined that baseline characteristics between the groups were not comparable despite frequency-based matching on age, gender, race/ethnicity. A propensity score analytic method was used to make the groups more comparable at baseline. The participant numbers are based on this model (218, 227) to account for baseline differences.
Measure: Count of Participants; unit: Participants
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized)
Number analyzed (Participants) | 218 | 227
Participants
  Hospitalization | 59 | 53
  Emergency Department | 43 | 51
  Urgent Care | 10 | 26

2. Secondary Outcome: Health Status and Quality of Life as Assessed by the Short Form-12 Question Physical Component Summary (SF-12 PCS) and the Short Form-12 Mental Component Summary (SF-12 MCS).
Description: Investigators will use the Short Form-12 question Physical Component Summary (SF-12 PCS) and the Short Form-12 Mental component Summary (SF-12 MCS) to measure physical and mental health status. Summary scores range from 0-100, with higher scores indicating a better self-reported level of health.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized)
Number analyzed (Participants) | 222 | 234
units on a scale
  SF-12 MCS Baseline | 49.0 [43.5 to 54.4] | 50.8 [45.5 to 56.2]
  SF-12 MCS 6 months | 51.2 [45.6 to 56.8] | 50.7 [45.2 to 56.1]
  SF-12 MCS 12 months | 50.1 [44.5 to 55.7] | 51.1 [45.7 to 56.5]
  SF-12 PCS Baseline | 35.5 [30.9 to 40.1] | 41.3 [36.8 to 45.8]
  SF-12 PCS 6 months | 35.6 [30.8 to 40.4] | 40.6 [36.0 to 45.1]
  SF-12 PCS 12 months | 36.4 [31.6 to 41.2] | 40.8 [36.3 to 45.4]

3. Secondary Outcome: Depressive Symptoms as Assessed by the 10 Item Version of the Center of Epidemiologic Studies-Depression Scale
Description: Investigators will use the 10 item version of the Center of Epidemiologic Studies-Depression scale to assess depressive symptoms. The possible range of scores is 0 to 10, with a score of zero indicating no depressive symptoms and a score of 10 indicating the most depressive symptoms
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized)
Number analyzed (Participants) | 222 | 234
units on a scale
  CES-D-10 Baseline | 3.82 [3.42 to 4.22] | 3.71 [3.33 to 4.09]
  CES-D-10 6 months | 3.49 [3.06 to 3.91] | 3.17 [2.79 to 3.56]
  CES-D-10 12 months | 3.48 [3.05 to 3.92] | 3.34 [2.94 to 3.73]

4. Secondary Outcome: Anxiety Symptoms as Assessed by the 5-item Version of the Geriatric Anxiety Inventory Short Form
Description: Investigators will use the 5-item version of the Geriatric Anxiety Inventory Short Form to measure anxiety symptoms. The scale is 0 to 5, with 0 points indicating zero anxiety symptoms and 5 indicating the most anxiety symptoms.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized)
Number analyzed (Participants) | 222 | 234
units on a scale
  Anxiety Index (0-5) Baseline | 1.80 [1.19 to 2.41] | 1.59 [0.99 to 2.19]
  Anxiety Index (0-5) 6 months | 1.51 [0.89 to 2.13] | 1.28 [0.68 to 1.88]
  Anxiety Index (0-5) 12 Months | 1.82 [1.20 to 2.45] | 1.29 [0.68 to 1.90]

5. Secondary Outcome: Loneliness as Assessed by the Short Scale for Measuring Loneliness in a Large Survey
Description: Investigators will use the Short Scale for Measuring Loneliness in a large survey. Three item measure with a three-point response scale from 1-3, with a score of 1 indicating the least loneliness and a score of 3 indicating the most loneliness.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized)
Number analyzed (Participants) | 222 | 234
units on a scale
  Loneliness (1-3) baseline | 1.70 [1.49 to 1.92] | 1.54 [1.33 to 1.76]
  Loneliness (1-3) 6 months | 1.66 [1.44 to 1.89] | 1.52 [1.30 to 1.73]
  Loneliness (1-3) 12 months | 1.75 [1.53 to 1.98] | 1.55 [1.33 to 1.77]

6. Secondary Outcome: Self-Efficacy as Assessed by the General Self-efficacy Scale to Measure an Individual's Sense of Perceived Self-efficacy.
Description: Investigators will use the General Self-efficacy Scale to measure an individual's sense of perceived self-efficacy. The total score ranges between 1 and 4, with 1 indicating low self-efficacy and 4 indicating high self-efficacy.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized)
Number analyzed (Participants) | 222 | 234
units on a scale
  Self-Efficacy (1-4) Baseline | 3.27 [3.19 to 3.35] | 3.44 [3.36 to 3.51]
  Self-Efficacy (1-4) 6 Months | 3.24 [3.15 to 3.32] | 3.35 [3.27 to 3.43]
  Self-Efficacy (1-4) 12 Months | 3.20 [3.11 to 3.28] | 3.29 [3.21 to 3.36]

7. Secondary Outcome: Resilience as Assessed by the Brief Resilience Scale
Description: Investigators will use the Brief Resilience Scale to measure the ability of individuals to bounce back from stress. Six item scale scored from 1-5, with a score of 1 indicating low resilience and a score of 5 indicating high resilience.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized)
Number analyzed (Participants) | 222 | 234
units on a scale
  Resilience (1-5) Baseline | 3.47 [3.25 to 3.70] | 3.60 [3.38 to 3.81]
  Resilience (1-5) 6 Months | 3.46 [3.22 to 3.70] | 3.49 [3.26 to 3.71]
  Resilience (1-5) 12 Months | 3.29 [3.05 to 3.52] | 3.64 [3.42 to 3.87]

8. Secondary Outcome: Social Support as Assessed by the 8-item Medical Outcomes Study Social Support Survey
Description: Investigators will use the 8-item medical outcomes study social support survey to measure social support. Scored from 1-5, and a score of 1 indicates lower levels of social support while a score of 5 indicates higher levels of social support.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized)
Number analyzed (Participants) | 222 | 234
units on a scale
  Social Support (1-5) Baseline | 3.48 [2.75 to 4.22] | 3.763 [2.9 to 4.36]
  Social Support (1-5) 6 Months | 3.50 [2.75 to 4.24] | 3.57 [2.84 to 4.30]
  Social Support (1-5) 12 Months | 3.54 [2.80 to 4.28] | 3.74 [3.01 to 4.47]

9. Secondary Outcome: Mobility Disability as Assessed by the Rosow-Breslow Scale
Description: The Rosow-Breslow scale is a composite measure of mobility disability. The composite score ranges from 0 to 3 with higher scores indicating greater disability.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized)
Number analyzed (Participants) | 222 | 234
units on a scale
  Rosow-Breslow (0-3) Baseline | 1.85 [1.61 to 2.10] | 1.45 [1.22 to 1.69]
  Rosow-Breslow (0-3) 6 Months | 1.69 [1.44 to 1.94] | 1.24 [1.01 to 1.48]
  Rosow-Breslow (0-3) 12 Months | 1.90 [1.65 to 2.16] | 1.47 [1.23 to 1.71]

10. Secondary Outcome: Physical Health as Assessed by the NAGI Test
Description: The NAGI test is a nine-item instrument scored from 1-5, with higher scores indicating less physical health.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized)
Number analyzed (Participants) | 222 | 234
units on a scale
  NAGI (0-5) Baseline | 3.02 [2.77 to 3.26] | 2.39 [2.16 to 2.62]
  NAGI (0-5) 6 Months | 2.74 [2.48 to 3.00] | 2.08 [1.85 to 2.32]
  NAGI (0-5) 12 Months | 2.97 [2.71 to 3.24] | 2.26 [2.02 to 2.50]

11. Secondary Outcome: Medical Conditions as Assessed by the Medical Conditions Questionnaire (MCQ)
Description: Medical Conditions Questionnaire has 9 yes/no questions on whether or not participants have ever had a condition like heart disease, cancer, diabetes, etc. It ranges from 0 to 9, with 0 indicating better overall health and 9 indicating poor overall health.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized)
Number analyzed (Participants) | 222 | 234
units on a scale
  MCQ Total (0-9) Baseline | 2.19 [2.02 to 2.37] | 2.10 [1.93 to 2.27]
  MCQ Total (0-9) 6 Months | 2.10 [1.92 to 2.29] | 1.70 [1.53 to 1.88]
  MCQ Total (0-9) 12 Months | 2.24 [2.05 to 2.43] | 1.88 [1.70 to 2.06]

ADVERSE EVENTS:
Time Frame: 12 months
Description: No adverser events were observed over the 12-month study period.
Arm/Group | Peer-to-peer Support (Non-randomized) | Standard Services (Non-randomized)
All-Cause Mortality (participants affected / at risk) | 0/222 | 0/234
Serious Adverse Events (participants affected / at risk) | 0/222 | 0/234
Other Adverse Events (participants affected / at risk) | 0/222 | 0/234

LIMITATIONS AND CAVEATS:
Our study was limited by the fact that we could not randomize participants and our groups were significantly different in some baseline characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT02308696/SAP_000.pdf
  • Study Protocol (2016-04-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT02308696/Prot_001.pdf